CLINICAL TRIAL: NCT06725420
Title: Comparison of the Effectiveness of Ultrasound-guided Local Steroid Injection vs Intramuscular Steroid Injection in the Treatment of Carpal Tunnel Syndrome: A Prospective, Randomized, Controlled, Single-blind Study
Brief Title: Ultrasound-Guided Injection vs Intramuscular Steroid for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Yılmaz, MD, Associate Professor (MD), S.B. Konya Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2023/1075
Record Dates: First submitted 2024-12-01; First posted 2024-12-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome (CTS); Chronic Pain
Keywords: Carpal tunnel syndrome; pain; Injection approach; Rehabilitation; Ultrasound-guided; Splints
MeSH Terms: conditions — Carpal Tunnel Syndrome; Chronic Pain; Pain | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- local steroid injection (Experimental): The group of patients who were injected with ultrasound-guided in-plane steroid and local anesthetic injection + wrist splint
  Interventions: Other: Ultrasound-guided local Injection; Device: Splinting
- intramuscular steroid injection (Experimental): The group of patients who received an intramuscular (gluteal) steroid and local anesthetic injection + wrist plint
  Interventions: Other: Intramuscular Steroid Injection; Device: Splinting
- Wrist splint (Experimental): The group of patients who received only a nighttime wrist splint
  Interventions: Device: Splinting

INTERVENTIONS:
Other: Ultrasound-guided local Injection — Ultrasound-Guided steroid injection and splinting in patients with carpal tunnel syndrome
  Other Names: wrist splint
  Arms: local steroid injection
Other: Intramuscular Steroid Injection — Intramuscular gluteal steroid injection and Splinting in Patients With Carpal Tunnel Syndrome
  Other Names: wrist splint
  Arms: intramuscular steroid injection
Device: Splinting — wrist night splint

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common and disability-causing entrapment neuropathy; however, a standardized protocol for first-line management has yet to be established. Different treatment approaches have their own positive and negative aspects.

The aim of this study is to compare the effectiveness of ultrasound-guided local steroid injection and intramuscular steroid injection in mild-to-moderate CTS. Patients will be assessed for pain levels, functional/symptom status, hand-finger strength, side effects, patient satisfaction, median nerve ultrasonographic measurements, and EMG before and after treatment .

DETAILED DESCRIPTION:
Patients evaluated through a detailed clinical examination and medical history review according to inclusion and exclusion criteria will provide written informed consent and will be assigned to one of three treatment groups using block randomization.

The patients' basic sociodemographic information (age, gender, body mass index, employment status, education level, marital status) and clinical data (dominant hand, duration of symptoms, comorbidities, hand to be treated, Tinel's/Phalen's sign, sleep quality, pain intensity, electrophysiological parameters.) will be recorded.

The first group (local steroid) will receive an ultrasound-guided local steroid injection (1 ml of 40 mg triamcinolone + 1 ml lidocaine) along with a nighttime wrist splint. The second group (intramuscular steroid) will receive a gluteal intramuscular injection (1 ml of 40 mg triamcinolone + 1 ml lidocaine) along with a nighttime wrist splint. The third group will receive only a nighttime wrist splint. All patients in the study groups were provided with prefabricated volar wrist splints to be used at night and, whenever possible, during the day for 2-3 hours. No medication or exercise therapy will be given to the patients.

All groups were evaluated based on examination findings (Tinel's/Phalen's test), pain intensity (VAS day and VAS night), hand grip strength (HGS), finger pinch strength (FGS), the Turkish version of the Boston Carpal Tunnel Questionnaire scores, sleep quality, the patient's subjective impression of improvement (satisfaction), electrophysiological parameters (two times), and ultrasound measurements (cross-sectional areas [CSA] and flattening ratio [long diameter/short diameter]) at the proximal inlet of the median nerve (at the level of the scaphoid and pisiform bones, at the level of the distal wrist crease) before treatment (baseline), at the end of treatment (two weeks), and six weeks after treatment. The evaluation parameters/outcomes will be made by the same researcher blind to the groups.

Patients will be questioned about undesirable effects at the end of the 2nd and 6th weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of typical CTS symptoms (numbness, tingling, paresthesias, or pain that may be provoked by nighttime or activity-related posture
* VAS score of ≥ 3/10
* Symptom duration longer than 12 weeks
* Positive Tinel's and/or Phalen's sign
* Electrophysiologically mild or moderate CTS being diagnosed.
* Volunteer to participate in study

Exclusion Criteria:

* Patients with shoulder, elbow, wrist, or finger problems (e.g., impingement syndrome, epicondylitis, history of fractures in the wrist, de Quervain's tenosynovitis, trigger finger, Complex Regional Pain Syndrome (CRPS), Dupuytren's contracture).
* Patients with a history of trauma or surgery in the affected hand, or those with significant anatomical deformities.
* Patients with systemic diseases such as rheumatological disorders, hypothyroidism, amyloidosis, diabetes, gout, or chronic kidney failure.
* Patients with conditions that may mimic CTS, such as polyneuropathy, plexopathy, cervical radiculopathy, or thoracic outlet syndrome.
* Patients with cognitive dysfunction or communication issues.
* Patients with severe CTS, neurological deficits (e.g., thenar atrophy, muscle weakness in thumb abduction/opposition), or those requiring surgical intervention.
* Patients who have received local steroid injections or physical therapy to the hand/wrist within the last 6 months.
* Patients who are receiving or will receive another/additional treatment for CTS.
* Pregnant or lactating women.
* Patients with active malignancies or local/systemic infections.
* Patients who are receiving any active treatment (e.g., NSAIDs, oral/intramuscular steroids, acupuncture, other pain medications).
* Patients with upper extremity involvement due to first motor neuron damage (e.g., stroke-hemiplegia, tetraparesis, multiple sclerosis).
* Patients with a bifid median nerve, persistent median artery, ganglion cyst, tenosynovitis, or tendinitis in the wrist.
* Use of a wrist splint during the last 6 months.
* Allergy to corticosteroids or local anesthetics, and blood diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
VAS pain | baseline, week 2 and week 6
  VAS pain day and night: 0 no pain; 10 unbearable/max. pain.
The Boston Carpal Tunnel Syndrome Questionnaire | baseline, week 2 and week 6
  The Turkish version of the Boston Carpal Tunnel Questionnaire score. It is used to evaluate the symptom severity and functionality of the patients. BCTQ is a questionnaire consisting of 2 parts: symptom severity scale (SSS) and functional status scale (FSS). Each item in both sections has 5 different answers that score between 1 and 5. The mean score is obtained by dividing the total score by the number of questions and ranges from 1 to 5, with a higher score indicating severe symptom.
Undesirable effects | Immediately, week 2 and week 6
  Possible side effects such as nerve/vessel injury, bleeding, skin discoloration, fat atrophy, infection, allergy, steroid exacerbation (transient pain starting 24 hours after the injection and lasting a few days), hypertension, and steroid-induced edema will be questioned and recorded in the patients

SECONDARY OUTCOMES:
Hand grip strength | baseline, week 2 and week 6
  Hand Grip Strength (HGS):
  Following the definitions outlined in the literature, HGS will be measured using Jamar hand dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Finger pinch strength | baseline, week 2 and week 6
  Finger Pinch Strength (FGS):
  Following the definitions outlined in the literature, FGS will be measured using Baseline pinch dynamometers. The patients will be asked to squeeze the dynamometer three times with maximum strength, allowing 30-60 seconds of rest between each attempt. The average force (in pounds/kg) will then be recorded.
Ultrasonographic evaluation of the median nerve | baseline, week 2 and week 6
  Ultrasonographic evaluation of the median nerve will be performed with a LA2-14A transducer /superficial linear probe (Samsung).
  The cross-sectional areas (CSA) of the median nerve at the proximal inlet of the carpal tunnel will be recorded. To identify the entrance of the carpal tunnel, measurements will be taken at the level of the distal wrist crease, at the scaphoid and pisiform bones. The assessments were conducted with the patients seated, facing the clinician, with their elbow bent at approximately 90˚, forearm in a supine position, and fingers in a semiflexed posture. Measurements were obtained using the manual tracing feature of the ultrasound device, excluding the hyperechoic nerve sheathThe CSA (mm2) will be determined. The average of the three measurements will be recorded.
Ultrasonographic evaluation of the median nerve | baseline, week 2 and week 6
  Ultrasonographic evaluation of the median nerve will be performed with a LA2-14A transducer /superficial linear probe (Samsung).
  The flattening ratio (long diameter/short diameter) of the median nerve at the proximal inlet of the carpal tunnel will be recorded. To identify the entrance of the carpal tunnel, measurements will be taken at the level of the distal wrist crease, at the scaphoid and pisiform bones. The assessments were conducted with the patients seated, facing the clinician, with their elbow bent at approximately 90˚, forearm in a supine position, and fingers in a semiflexed posture. Measurements were obtained using the manual tracing feature of the ultrasound device, flattening ratio will be determined. The average of the three measurements will be recorded.
Sleep quality | Baseline, week 2 and week 6
  Sleep quality was evaluated using a single 4-point (0 = very bad, 3 = very good) Likert-type question from item 6 of the Pittsburgh Sleep Quality Index
Electrophysiological (nerve conduction) parameters | baseline and week 6
  Electrophysiological parameters (median nerve distal motor latency) will be measured at two time points (baseline and week 6).
Electrophysiological (nerve conduction) parameters | baseline and week 6
  Electrophysiological (nerve conduction) parameters (median sensory nerve distal latency) will be measured at two time points (baseline and week 6).
Electrophysiological (nerve conduction) parameters | baseline and week 6
  Electrophysiological parameters (sensory and motor nerve conduction velocities) will be measured at two time points (baseline and week 6).
Electrophysiological (nerve conduction) parameters | baseline and week 6
  Electrophysiological parameters (amplitudes of compound muscle action potential and sensory nerve action potential) will be measured at two time points (baseline and week 6).
Patient satisfaction | baseline, week 2 and week 6
  Patient satisfaction (Subjective impression of improvement):
  Satisfaction levels of patients will be questioned. In the assessment consisting of five clauses with Likert-type scales, the clauses will be described as follows: 1, 'no satisfaction at all'; 2, 'no satisfaction'; 3, neutral (no positive or negative effect); 4, 'satisfied'; and 5, 'very satisfied'.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No